CLINICAL TRIAL: NCT03978871
Title: Effect of Emotion Mindsets on Emotion Processing: A Multilevel Experimental Investigation
Brief Title: Effect of Emotion Mindsets on Emotion Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Auburn University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18021; R21HD097537 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Emotions
Keywords: Brain; Functional Neuroimaging; Stress, Psychological; Emotions; Psychology, Developmental
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth Mindset (Experimental): Persuasive education about emotions, brain development, and teenagers' ability to learn how to manage emotions
  Interventions: Behavioral: Growth Mindset
- Brain Education (Active Comparator): Neutral education about functions of different parts of the brain
  Interventions: Behavioral: Brain Education

INTERVENTIONS:
Behavioral: Growth Mindset — Growth emotion mindset induction
  Arms: Growth Mindset
Behavioral: Brain Education — Brain education
  Arms: Brain Education

SUMMARY:
The guiding scientific premise for this research is that a growth emotion mindset will promote more adaptive emotion processing than a fixed emotion mindset. Because emotional sensitivity is particularly salient in adolescent girls, we will focus on this group. Using an experimental design, adolescent girls will be randomly assigned to either a mindset manipulation or a control group (brain education). Each group will complete a 25-minute computer-based lesson followed by a social stressor and a functional magnetic resonance imaging session. Two specific aims will be addressed: (1) to determine whether a growth mindset induction, relative to a control condition, predicts more adaptive emotion processing at the neural, behavioral, and psychological levels of processing; and (2) to determine whether neural processing of emotion accounts for the effect of a growth emotion mindset manipulation on behavioral and psychological processing of emotion. This study builds on a strong empirical database establishing the effect of mindsets on multiple domains of functioning but will be the first to examine the implications of a growth vs. fixed mindset about emotion for emotion processing in adolescent girls, thereby elucidating one specific youth attribute that can support or disrupt emotional development.

DETAILED DESCRIPTION:
150 adolescent girls will complete baseline measures and then be randomly assigned to one of two conditions and will complete a computer-based lesson (see below). Girls will then engage in a social stressor outside of the scanner as well as an emotional challenge and cognitive control task in the scanner and will complete post-scan measures. Two and four months after the scan session they will complete additional survey measures.

Experimental condition: The (Growth Emotion Mindset) GEM manipulation, involves 6 components: (1) Introduction: discussion of emotional experiences in teenagers; (2) Explanation of neuroplasticity, emphasizing the potential for changes in the brain and modification of emotions during adolescence; (3) Scientific evidence for the effect of emotion regulation training on mood improvement; (4) Brief factual quizzes and written summary of key points; (5) Scenarios in which older youth describe challenging situations when they used growth mindsets to help regulate negative emotions; and (6) Self-persuasion exercise: a. Girls read a hypothetical scenario about an emotional challenge and describe their likely thoughts and feelings; b. Girls imagine the same event happening to another (younger) teen and help them understand how they can change, integrating what they learned about malleability of the brain and emotion.

Control condition: The control condition involves a structurally similar session, with the same number and type of reading and writing activities, that focuses on general education about the brain.

Social stressor. Using an adapted version of the Trier Social Stressor Test, girls will prepare a speech in which they convince a group of peers (who ostensibly will watch a video of the speech; in reality, there are no peers) that they should be selected for a fictional television show about teens' ability to form friendships. Girls face a computer screen displaying their image while preparing and presenting a speech. At intervals of 20 seconds, a female evaluator will mark a clipboard. Before and after the Trier, girls will rate several dimensions of state negative affect. After the Trier, girls will rate their use of in vivo emotion regulation strategies.

Girls will then undergo scanner training and watch a neutral video during an anatomical scan.

Emotional challenge (Social Evaluation Task). Girls will watch validated videos created for functional magnetic resonance imaging, which depict females making one of three types of statements with matching affective expression: negative social-evaluative, positive social-evaluative, or neutral. Before each video, girls will receive a prompt instructing them to imagine how they would feel if the female were a friend and if the statement was directed either toward the participant (immerse), or toward a stranger (reframe). After the cue, there will be a pause, presentation of the video, and another pause. After each trial, the participant will rate how bad they feel on a 5-point scale.

Resting state. Following the emotional challenge, girls will remain still and fixate on a central cross. Greater ability to flexibly engage and disengage emotion regulation in response to changing external challenges (imposed by negative, positive, and neutral videos) is expected to be reflected in the functional connectome for minutes beyond the emotional challenge task, resulting in more within-network connectivity in cognitive control networks as well as increased connectivity with emotion regions in girls engaged in proactive emotion regulation.

Emotional go-nogo. This task combines a cognitive control task (go-nogo) with emotion distractors depicting negative (social rejection), positive (social acceptance), or neutral (scrambled) images taken from a validated set of stimuli. Letters are presented sequentially in a small box at the center of the screen, with emotion distractors in the background. The distractors are presented alone , prior to presentation of the letter, to make it difficult to ignore the emotional content. Girls are instructed to ignore the images and respond as quickly as possible without sacrificing accuracy with a button press to every letter (go trials), except for Xs (no-go; 25 percent of trials). Girls acquire a prepotent tendency to press and must inhibit their responses during X trials.

Edited June 2020:

Anticipated 75% and 100% enrollment dates as well as primary and final study completion dates and primary endpoint analyses and reporting of results were changed due to recruitment and data collection obstacles posed by the coronavirus pandemic. The new dates were estimated based on the assumption that some recruitment and data collection will resume in the fall of 2020. If this is not possible or if families are reluctant to complete sessions, completion dates may need to be changed again at a later date.

Edited November 2021:

Although the 75% enrollment was reached, anticipated 100% enrollment date as well as primary and final study completion dates and primary endpoint analyses and reporting of results were changed due to ongoing recruitment and data collection obstacles posed by the coronavirus pandemic. Although a small amount of recruitment and data collection resumed fall of 2020-fall of 2021, obstacles still remain due to school and family reluctance to participate in research.

ELIGIBILITY:
Inclusion Criteria:

* Female age 13-18 years old
* Over-sample (approximately 1/3 of sample) for score >= .75 standard deviation (SD) on a screening measure of fixed mindset about emotion
* English-speaking
* Ability to independently complete tasks and measures

Exclusion Criteria:

* History of surgery involving metal implants
* Possible metal fragments in the eyes or other parts of body
* Pacemaker
* A history of claustrophobia
* Braces
* Weighing over 250 pounds
* Pregnancy or possibility of being pregnant
* Severe medical conditions (e.g., blind or deaf, head trauma)
* Learning disability or other condition that interferes with ability to complete tasks

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Identify as female
Enrollment: 163 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen D Rudolph, PhD, Principal Investigator — University of Illinois, Urbana Champaign
Locations (1):
- University of Illinois, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share our behavioral data publicly on the Open Science Framework upon publication. De-identified neuroimaging data will be organized according to the Brain Imaging Data Structure (BIDS) guidelines, a standard developed to provide a consistent framework for storing and sharing neuroimaging data. These data will then be shared on the openfMRI platform https://openfmri.org upon publication.
Time Frame: Upon publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from local high schools between August of 2018 and June of 2022. The first participant was enrolled in the main study in August of 2018 and the last participant was enrolled in June of 2022. The study was completed by October of 2022.
Pre-assignment Details: One additional participant consented, but then declined participation due to concerns about claustrophobia while in the fMRI machine.
Groups:
- Brain Education: Neutral education about functions of different parts of the brain
  Control: Brain education
Period: Overall Study
Arm/Group | Growth Mindset | Brain Education
Started | 81 | 82
2-Month Follow-up | 72 | 75
4-Month Follow-up | 74 | 75
Completed | 70 | 70
Not Completed | 11 | 12
Not completed — Lost to Follow-up | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Mindset | Brain Education | Total
Number analyzed (Participants) | 81 | 82 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 81 | 82 | 163
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.63 (1.10) | 15.72 (1.06) | 15.68 (1.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 82 | 163
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 7 | 10 | 17
  Asian | 8 | 6 | 14
  Latina/o | 4 | 3 | 7
  White | 52 | 56 | 108
  Other | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 81 | 82 | 163
Grade [Count of Participants; unit: Participants]
  Eighth Grade | 6 | 10 | 16
  Ninth Grade | 38 | 29 | 67
  Tenth Grade | 20 | 25 | 45
  Eleventh Grade | 14 | 17 | 31
  Twelfth Grade | 3 | 1 | 4
Marital Status of Caregiver [Count of Participants; unit: Participants] — Population: one participant did not fill out this information.
  Participants
    Married: number analyzed (Participants) | 81 | 81 | 162
    Married | 62 | 63 | 125
    Single (never married): number analyzed (Participants) | 81 | 81 | 162
    Single (never married) | 6 | 7 | 13
    Single (divorced): number analyzed (Participants) | 81 | 81 | 162
    Single (divorced) | 11 | 8 | 19
    Separated: number analyzed (Participants) | 81 | 81 | 162
    Separated | 1 | 1 | 2
    Other (specified): number analyzed (Participants) | 81 | 81 | 162
    Other (specified) | 1 | 2 | 3
Total Gross Annual Family Income [Count of Participants; unit: Participants] — Total family income was assessed on a 7-point scale.
  Participants
    $15-29,999 | 5 | 3 | 8
    $30-44,999 | 7 | 7 | 14
    $45-59,999 | 15 | 8 | 23
    $60-74,999 | 9 | 6 | 15
    $75-89,999 | 4 | 5 | 9
    $90,000 and over | 40 | 50 | 90
    $0-14,999 | 0 | 2 | 2
    Missing | 1 | 1 | 2
Female Caregiver's Highest Level of Education [Count of Participants; unit: Participants]
  Professional Degree (M.D., PhD., etc.) | 7 | 6 | 13
  Master's Degree (M.A., M.S.) | 19 | 23 | 42
  Some graduate school | 6 | 6 | 12
  Bachelor's degree (B.A., B.S.) | 25 | 20 | 45
  Associate's degree | 4 | 7 | 11
  Some college | 10 | 15 | 25
  High school diploma | 8 | 4 | 12
  Missing | 1 | 1 | 2
  Some high school | 1 | 0 | 1
Male Caregiver's Highest Level of Education [Count of Participants; unit: Participants]
  Professional Degree (M.D., PhD., etc.) | 12 | 17 | 29
  Master's Degree (M.A., M.S.) | 15 | 11 | 26
  Bachelor's Degree (B.A., B.S.) | 16 | 18 | 34
  Associate's Degree | 8 | 9 | 17
  Some college | 12 | 10 | 22
  High school diploma | 5 | 0 | 5
  Some high school | 1 | 0 | 1
  Missing | 12 | 13 | 25
  Some graduate school | 0 | 3 | 3
  8th grade completed | 0 | 1 | 1
Caregiver 1 Relationship to Child [Count of Participants; unit: Participants]
  Biological Mother | 69 | 70 | 139
  Stepmother | 1 | 1 | 2
  Biological Father | 9 | 9 | 18
  Other | 2 | 1 | 3
  Missing | 0 | 1 | 1
Caregiver 2 Relationship to Child [Count of Participants; unit: Participants]
  Biological Father | 55 | 53 | 108
  Stepfather | 2 | 3 | 5
  Biological Mother | 8 | 10 | 18
  Other | 3 | 1 | 4
  Missing | 13 | 14 | 27
  Stepmother | 0 | 1 | 1
Risk Group [Count of Participants; unit: Participants] — Participants were identified as being at high or low risk for negative emotionality based on their initial levels of low/average fixed mindsets vs. high fixed mindsets,
  Participants
    Low Risk | 54 | 54 | 108
    High Risk | 27 | 28 | 55
School Code [Count of Participants; unit: Participants]
  School 1 | 3 | 6 | 9
  School 2 | 7 | 5 | 12
  School 3 | 1 | 0 | 1
  School 4 | 4 | 2 | 6
  School 5 | 2 | 8 | 10
  School 6 | 16 | 2 | 18
  School 7 | 7 | 21 | 28
  School 8 | 12 | 2 | 14
  School 9 | 1 | 8 | 9
  School 10 | 3 | 7 | 10
  School 11 | 1 | 4 | 5
  School 12 | 12 | 6 | 18
  School 13 | 5 | 1 | 6
  School 14 | 2 | 3 | 5
  School 15 | 5 | 7 | 12
Emotion Mindset Scale (Pre-Induction EMS) [Mean (Standard Deviation); unit: score on a scale] — Participants completed a six-item fixed emotion mindset measure (EMS-fixed) measure, prior to the induction lessons (pre-induction EMS). Items were drawn from the Implicit Theories of Emotion Scale (Tamir et al., 2007) and the Emotion Mindset Scale (EMS; Livingstone, 2013). Participants rated each item on a 6-point scale (1 = Strongly Disagree to 6 =Strongly Agree). Means were computed for these items, with higher scores representing a higher fixed emotion mindset mindset. Minimum=1 Maximum=6 High= more fixed emotion mindset, worse outcome.
  score on a scale | 3.03 (0.96) | 3.03 (0.92) | 3.03 (0.94)
Emotion Mindset Scale (Post-Induction EMS) [Mean (Standard Deviation); unit: score on a scale] — Participants completed a six-item fixed emotion mindset measure (EMS-fixed) measure, following the induction lessons (post-induction EMS). Items were drawn from the Implicit Theories of Emotion Scale (Tamir et al., 2007) and the Emotion Mindset Scale (EMS; Livingstone, 2013). Participants rated each item on a 6-point scale (1 = Strongly Disagree to 6 =Strongly Agree). Means were computed for these items, with higher scores representing a higher fixed emotion mindset mindset. Minimum=1 Maximum=6 High= more fixed emotion mindset, worse outcome..
  score on a scale | 2.17 (0.90) | 2.76 (0.90) | 2.46 (0.95)
Emotion Regulation Self-Efficacy (Pre-ESES) [Mean (Standard Deviation); unit: score on a scale] — Participants completed a measure assessing their perceived ability to manage emotions prior to the induction. Items were derived from the using and managing your own emotions subscale of the Youth-ESES (5 items; Qualter et al., 2015). Participants rated the items on a 5-point Likert scale (1 = Disagree Strongly to 5 = Agree Strongly). Scores were computed as the mean of the items, with higher scores indicating greater emotion regulation self-efficacy. Population: One participant did not fully complete this measure.
  score on a scale
    number analyzed (Participants) | 80 | 82 | 162
    (all) | 3.53 (0.79) | 3.34 (0.89) | 3.43 (0.84)
Emotion Regulation Self-Efficacy (Post-ESES) [Mean (Standard Deviation); unit: score on a scale] — Participants completed a measure assessing their perceived ability to manage emotions following the induction. Items were derived from the using and managing your own emotions subscale of the Youth-ESES (5 items; Qualter et al., 2015). Participants rated the items on a 5-point Likert scale (1 = Disagree Strongly to 5 = Agree Strongly). Scores were computed as the mean of the items, with higher scores indicating greater emotion regulation self-efficacy.This measure assesses participants' levels of self-efficacy post-induction condition.
  score on a scale | 3.79 (0.82) | 3.40 (0.86) | 3.59 (0.86)
Tamir pre self-efficacy [Mean (Standard Deviation); unit: score on a scale] — To assess emotion regulation self-efficacy participants completed a self-efficacy measure adapted from Tamir and colleagues (2007). Prior to the induction, participants were asked to rate 12 emotion-eliciting events drawn from daily life. Three scenarios were adapted from the Tamir self-efficacy measure (Tamir et al. 2007. Participants rated how confident they were in their ability to control their emotions in each scenario on a 5-point scale (1 = Not at All to 5 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting greater self-efficacy.
  score on a scale | 2.89 (0.62) | 2.70 (0.62) | 2.79 (0.63)
Tamir post self-efficacy [Mean (Standard Deviation); unit: score on a scale] — To assess emotion regulation self-efficacy participants completed a self-efficacy measure adapted from Tamir and colleagues (2007). Following the induction, participants were asked to rate 12 emotion-eliciting events drawn from daily life. Participants rated how confident they were in their ability to control their emotions in each scenario on a 5-point scale (1 = Not at All to 5 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting greater self-efficacy.This measure assesses participants' levels of self-efficacy post-induction condition.
  score on a scale | 3.16 (0.67) | 2.72 (0.70) | 2.94 (0.72)
Youth Emotion Regulation and Dysregulation Scale (YERD) [Mean (Standard Deviation); unit: score on a scale] — To assess emotion (dys)regulation, participants completed a novel 44-item emotion regulation measure. Items were rated on a 5-point scale (1 = Not at All to 5 = Very Much). Factor analyses yielded three emotion regulation strategies factors- proactive engagement, involuntary dysregulation, and disengagement. Scores were computed as the mean of the items on each factor (1 = Not at All to 5 = Very Much), with higher scores reflecting higher levels of response. Higher scores on proactive engagement are adaptive and higher scores on involuntary dysregulation and disengagement are maladaptive.
  score on a scale
    Proactive Engagement Factor | 2.96 (0.77) | 2.70 (0.77) | 2.83 (0.78)
    Involuntary Dysregulation Factor | 2.44 (0.66) | 2.47 (0.75) | 2.45 (0.71)
    Disengagement Factor | 3.23 (0.65) | 3.02 (0.73) | 3.13 (0.69)
Emotion Regulation Strategies (ERS) [Mean (Standard Deviation); unit: score on a scale] — Participants completed a measure to assess the emotion regulation strategies (ERS) they used during the Trier Social Stress Test (TSST). Items were rated on a 5-point scale (1 = Not at All to 5 = Very Much). Factor analyses yielded three emotion regulation strategies factors- involuntary dysregulation, proactive engagement, and cognitive avoidance. Scores were computed as the mean of the items on each factor (1 = Not at All to 5 = Very Much). Higher scores on proactive engagement are considered adaptive and higher scores on involuntary dysregulation and cognitive avoidance are maladaptive. Population: Six participants refused to complete the Trier Social Stress Test so this measure did not apply to them.
  score on a scale
    Proactive engagement factor: number analyzed (Participants) | 77 | 80 | 157
    Proactive engagement factor | 3.05 (1.01) | 2.71 (1.02) | 2.87 (1.02)
    Involuntary dysregulation factor: number analyzed (Participants) | 77 | 80 | 157
    Involuntary dysregulation factor | 2.54 (1.01) | 2.75 (1.05) | 2.65 (1.03)
    Cognitive avoidance factor: number analyzed (Participants) | 77 | 80 | 157
    Cognitive avoidance factor | 2.77 (1.03) | 2.63 (1.00) | 2.70 (1.01)
Short Mood and Feelings Questionnaire (SMFQ) Child [Mean (Standard Deviation); unit: score on a scale] — Participants completed the short form of the Mood and Feelings Questionnaire (SMFQ; Angold et al., 1995) to assess depressive symptoms (13 items). The original version was modified (Liang & Eley, 2005) to provide a 4-point response format (1 = Not at All, 2 = A Little Bit, 3 = Pretty Much, 4 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting higher levels of depressive symptoms. Population: Two participants did not fully complete this measure.
  score on a scale
    number analyzed (Participants) | 80 | 81 | 161
    (all) | 1.84 (0.68) | 1.80 (0.64) | 1.82 (0.66)
Revised Child Manifest Anxiety Scale (RCMAS) [Mean (Standard Deviation); unit: score on a scale] — Participants completed the Revised Child Manifest Anxiety Scale (RCMAS; Reynolds & Richmond, 1985). The RCMAS includes 28 items assessing anxiety symptoms (e.g., "I often worry about something bad happening to me.") rated on a dichotomous scale (0 = No, 1 = Yes). Total anxiety scores were created by taking the sum of the items, with higher scores reflecting higher levels of anxiety. The RCMAS shows strong internal consistency (Reynolds & Richmond, 1978) and test-retest reliability (Wisniewski et al., 1987).
  score on a scale | 13.62 (6.08) | 13.61 (6.24) | 13.61 (6.14)
Affect Scale [Mean (Standard Deviation); unit: score on a scale] — Before (mt1pretrierneg) and after (mt1posttrierneg) completing the Trier Social Stress Test (TSST) at baseline, participants completed ratings of negative emotions (10 items), modified from another affect measure (Owens et al., 2019), to test the efficacy of the TSST. Participants rated their emotions on a 100-point scale (0 = Not at All to 100 = Extremely) to indicate the extent they were feeling a negative emotion at that particular moment. Scores were computed as the mean of the items on each subscale, with higher scores reflecting higher levels of negative emotions. Population: Some participants did not fully complete these measures.
  score on a scale
    mean Negative Affect pre trier (mt1pretrierneg) | 7.21 (9.68) | 7.90 (8.57) | 7.55 (9.12)
    mean Negative Affect post trier (mt1posttrierneg): number analyzed (Participants) | 77 | 80 | 157
    mean Negative Affect post trier (mt1posttrierneg) | 15.05 (14.83) | 16.51 (14.35) | 15.78 (14.56)
Induction Validity Check [Mean (Standard Deviation); unit: score on a scale] — To assess the equivalence of the emotion mindset and control conditions, participants completed a short questionnaire. Participants rated four items (interesting, informative, persuasive, and easy to understand) on a 10-point scale. To assess post-induction affect, participants rated their general emotional state on a 10-point scale (1 = Very Negative to 10 = Very Positive) Scores were computed as the mean of the items. This item was included as a separate variable in analyses, with higher scores indicating more positive affect post-induction.
  score on a scale
    mean induction validity (mt1validity) | 8.01 (1.30) | 7.21 (1.57) | 7.61 (1.49)
    Interesting (t1interesting) | 7.46 (1.79) | 7.05 (2.05) | 7.25 (1.93)
    Informative (t1informative) | 8.35 (1.61) | 8.01 (1.88) | 8.18 (1.75)
    Persuasive (t1persuasive) | 7.20 (2.02) | 5.55 (2.54) | 6.37 (2.43)
    Easy to Understand (t1understand) | 9.04 (1.62) | 8.22 (1.83) | 8.63 (1.77)
    Validity Affect (t1validityaffect) | 7.86 (1.83) | 7.23 (1.50) | 7.55 (1.70)
Social Evaluation (SET) Task [Mean (Standard Deviation); unit: units on a scale] — The Social Evaluation Task examines emotion reactivity with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative immerse or reframe), praise (positive immerse or reframe), or neutral statements (neutral immerse). In immerse trials, participants imagined that the person was a close friend. During the reframe trials, participants imagined that the person was an actor. After each trial, participants rated how they felt from 1 (Very Good) to 5 (Very Bad). Means of each condition were computed with higher scores indicating more negative emotions. Population: Some participants did not participate in this task and other participants' data was lost or not captured due to technological issues.
  units on a scale
    Mean Negative Immerse: number analyzed (Participants) | 74 | 76 | 150
    Mean Negative Immerse | 4.34 (0.51) | 4.28 (0.63) | 4.31 (0.57)
    Mean Negative Reframe: number analyzed (Participants) | 74 | 76 | 150
    Mean Negative Reframe | 3.49 (0.51) | 3.45 (0.67) | 3.48 (0.59)
    Mean Positive Immerse: number analyzed (Participants) | 74 | 76 | 150
    Mean Positive Immerse | 1.61 (0.60) | 1.61 (0.58) | 1.61 (0.59)
    Mean Positive Reframe: number analyzed (Participants) | 74 | 76 | 150
    Mean Positive Reframe | 2.39 (0.64) | 2.32 (0.60) | 2.36 (0.62)
    Mean Neutral Immerse: number analyzed (Participants) | 74 | 76 | 150
    Mean Neutral Immerse | 2.90 (0.33) | 2.87 (0.43) | 2.89 (0.38)
Socioemotional Go/No-go Task- Reaction Time [Mean (Standard Deviation); unit: Reaction time in milliseconds] — The socioemotional Go/No-go presents participants with a socially appetitive image, socially aversive image, or neutral image. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond as quickly as possible to every letter. Responses during these 500 ms were used for analysis. Mean reaction times (RT) in milliseconds to positive stimuli (pos.correctgoRT), negative stimuli (neg.correctgoRT) and neutral stimuli (neu.correctgoRT) were calculated, with higher numbers indicating slower RT and more attention to image content. Population: Some participants chose not to participate this task. The rest of the missing data is a result of scanner or technological issues or participant error.
  Reaction time in milliseconds
    mean reaction time to correct go positive condition (pos.correctgoRT): number analyzed (Participants) | 75 | 75 | 150
    mean reaction time to correct go positive condition (pos.correctgoRT) | 427.89 (38.25) | 433.44 (28.81) | 430.66 (33.86)
    mean reaction time to correct go negative condition (neg.correctgoRT): number analyzed (Participants) | 75 | 75 | 150
    mean reaction time to correct go negative condition (neg.correctgoRT) | 424.19 (36.18) | 431.78 (31.89) | 427.98 (34.20)
    mean reaction time to correct go neutral condition (neu.correctgoRT): number analyzed (Participants) | 74 | 75 | 149
    mean reaction time to correct go neutral condition (neu.correctgoRT) | 430.37 (33.42) | 434.35 (37.70) | 432.37 (30.63)
Socioemotional Go/No-go Task- Accuracy [Mean (Standard Deviation); unit: score on a scale] — The socioemotional Go/No-go presents participants with a socially appetitive image, socially aversive image, or neutral image. After, a letter was superimposed on the image. Participants were instructed to respond to every letter except for 'X'. Participants completed 4 blocks of each condition. Accurate responses to the letters after the socially appetitive images (positive accuracy), socially aversive image (negative accuracy) and neutral image (neutral accuracy) were indicated (0-1 scale). Mean scores across the four blocks were calculated, with higher scores indicating more accuracy. Population: Some participants chose not to participate this task. The rest of the missing data is a result of scanner or technological issues or participant error.
  score on a scale
    Positive accuracy: number analyzed (Participants) | 75 | 75 | 150
    Positive accuracy | 0.63 (0.10) | 0.60 (0.12) | 0.62 (0.11)
    negative accuracy: number analyzed (Participants) | 75 | 75 | 150
    negative accuracy | 0.64 (0.10) | 0.62 (0.12) | 0.63 (0.11)
    neutral accuracy: number analyzed (Participants) | 75 | 75 | 150
    neutral accuracy | 0.65 (0.11) | 0.63 (0.13) | 0.64 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Pre to Post Mindset Manipulation on Emotion Mindset Scale (Measures Beliefs About Whether Emotions Are Fixed or Malleable)
Description: Participants completed a six-item fixed emotion mindset measure (EMS-fixed) measure, prior to (pre-induction EMS) and following the induction lessons (post-induction EMS). Items were drawn from the Implicit Theories of Emotion Scale (Tamir et al., 2007) and the Emotion Mindset Scale (EMS; Livingstone, 2013). Participants rated each item on a 6-point scale (1 = Strongly Disagree to 6 =Strongly Agree). Means were computed for these items, with higher scores representing a higher fixed emotion mindset mindset. For this analysis, we compared mean change scores across the two conditions (mindset and control). Minimum=1 Maximum=6 High= more fixed emotion mindset, worse outcome
Time Frame: Pre vs. Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 81 | 82
score on a scale
  pre-induction EMS | 3.03 (0.96) | 3.03 (0.92)
  post-induction EMS | 2.17 (0.90) | 2.76 (0.90)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation). This is a test of between by within-subjects interaction effect; Test type: Superiority; p < 0.001, ANOVA — The threshold for statistical significance was p = 0.05; degrees of freedom =1

2. Primary Outcome: Mean Change From Pre to Post Mindset Manipulation on Emotional Self-efficacy Scale (Measure Beliefs About Ability to Control Emotions)
Description: Participants completed a measure assessing their perceived ability to manage emotions prior to and following the induction. Items were derived from the using and managing your own emotions subscale of the Youth-Emotional Self-efficacy Scale (5 items; Qualter et al., 2015). Participants rated the items on a 5-point Likert scale (1 = Disagree Strongly to 5 = Agree Strongly). Scores were computed as the mean of the items, with higher scores indicating greater emotion regulation self-efficacy. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome
Time Frame: Pre vs. Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 80 | 82
score on a scale
  pre-Emotional Self-efficacy | 3.53 (0.79) | 3.34 (0.89)
  post-Emotional Self-efficacy | 3.79 (0.82) | 3.40 (.86)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.023, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation). This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.034, ANCOVA; degrees of freedom = 1

3. Primary Outcome: Mean Change From Pre to Post Mindset Manipulation on Emotional Self-efficacy Vignettes (Measure Beliefs About Ability to Control Emotions in Specific Situations)
Description: To assess emotion regulation self-efficacy participants completed a self-efficacy measure adapted from Tamir and colleagues (2007). Prior to and following the induction, participants were asked to rate 12 emotion-eliciting events drawn from daily life. Three scenarios were adapted from the Tamir self-efficacy measure (Tamir et al. 2007. Participants rated how confident they were in their ability to control their emotions in each scenario on a 5-point scale (1 = Not at All to 5 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting greater self-efficacy. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome
Time Frame: Pre vs. Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 81 | 82
score on a scale
  pre-induction Emotional Self-Efficacy | 2.89 (0.62) | 2.70 (0.62)
  post-induction Emotional Self-Efficacy | 3.16 (0.67) | 2.72 (0.70)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The threshold for statistical significance was p = 0.0.5; p < .001, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; [analysis description as in outcome 2, analysis 2]; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.002, ANCOVA; degrees of freedom = 1

4. Primary Outcome: Mean Difference in Performance on Go/Nogo Task- Reaction Time
Description: The socioemotional Go/No-go presents participants with a socially appetitive image, socially aversive image, or neutral image. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond as quickly as possible to every letter. Responses during these 500 ms were used for analysis. Mean reaction times (RT) in milliseconds to positive stimuli (pos.correctgoRT), negative stimuli (neg.correctgoRT) and neutral stimuli (neu.correctgoRT) were calculated, with higher numbers indicating slower RT.
  Will compare mean performance as reflected in reaction time across the two conditions (mindset and control)
Time Frame: Post Mindset Manipulation: baseline
Population: 1 participant's data could not be used in the growth mindset condition in analyses. The means reported here for the growth mindset condition are slightly different than the means reported at baseline because here we are reporting the means of the participants analyzed, which does not include the one participant who's data could not be used.
Measure: Mean (Standard Deviation); unit: Reaction time in milliseconds
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 74 | 75
Reaction time in milliseconds
  positive correct_go reaction time | 427.40 (38.28) | 433.44 (28.81)
  negative correct_go reaction time | 423.37 (35.72) | 431.78 (31.89)
  neutral correct_go reaction time | 430.37 (33.42) | 434.35 (37.70)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education). This is a test of between-subjects effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.227, ANOVA; degrees of freedom = 1

5. Primary Outcome: Mean Difference in Performance on Go/Nogo Task- Accuracy
Description: The socioemotional Go/No-go presents participants with a socially appetitive image, socially aversive image, or neutral image. After, a letter was superimposed on the image. Participants were instructed to respond to every letter except for 'X'. Participants completed 4 blocks of each condition. Accurate responses to the letters after the socially appetitive images (positive accuracy), socially aversive image (negative accuracy) and neutral image (neutral accuracy) were indicated (0-1 scale). Mean scores across the four blocks were calculated, with higher scores indicating more accuracy. Will compare mean performance as reflected in accuracy across the two conditions (mindset and control)
Time Frame: Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 75 | 75
units on a scale
  positive accuracy | 0.63 (0.10) | 0.60 (0.12)
  negative accuracy | 0.64 (0.10) | 0.62 (0.12)
  neutral accuracy | 0.65 (0.11) | 0.63 (0.13)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect for accuracy (Growth Mindset vs. Brain Education). This is a test of between-subjects effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.272, ANOVA; degrees of freedom = 1

6. Primary Outcome: Mean Difference in Emotion Regulation Strategies on the Emotion Regulation Strategy Scale
Description: Participants completed a measure to assess the emotion regulation strategies (ERS) they used during the Trier Social Stress Test (TSST). Items were rated on a 5-point scale (1 = Not at All to 5 = Very Much). Factor analyses yielded three emotion regulation strategies factors- involuntary dysregulation, proactive engagement, and cognitive avoidance. Scores were computed as the mean of the items on each factor (1 = Not at All to 5 = Very Much), with higher scores reflecting higher levels of each type of response. In analyses, we compare mean scores for each of these factors across the two conditions (mindset and control). Higher scores on proactive engagement are considered adaptive and higher scores on involuntary dysregulation and cognitive avoidance are considered maladaptive.
Time Frame: Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 80 | 77
units on a scale
  involuntary dysregulation | 2.54 (1.01) | 2.75 (1.05)
  proactive engagement | 3.05 (1.01) | 2.71 (1.02)
  cognitive avoidance | 2.77 (1.03) | 2.63 (1.00)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) for the ERS emotion regulation involuntary dysregulation subscale post psycho-educational lesson. This is a test of between-subjects effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.217, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) for the ERS emotion regulation involuntary dysregulation subscale post psycho-educational lesson. This is a test of between-subjects effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.458, ANCOVA; degrees of freedom = 1
Statistical Analysis 3: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) for the ERS emotion regulation proactive engagement subscale post psycho-educational lesson. This is a test of between-subjects effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.037, ANOVA; degrees of freedom = 1
Statistical Analysis 4: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) for the ERS emotion regulation proactive engagement subscale post psycho-educational lesson. This is a test of between-subjects effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.107, ANCOVA; degrees of freedom = 1
Statistical Analysis 5: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) for the ERS emotion regulation cognitive avoidance subscale post psycho-educational lesson. This is a test of between-subjects test; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.369, ANOVA; degrees of freedom = 1

7. Primary Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Amygdala Activation- Social Evaluation Task
Description: The Social Evaluation Task (SET) examines emotion reactivity and regulation with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative condition), praise (positive condition) or neutral statements (neutral condition). Participants were asked to imagine the person was either an actor practicing lines (reframe condition), or a close friend (immerse condition). Participants were subsequently asked to rate how they felt on a 5 item Likert scale from "Very Good" to "Very Bad". To reduce the influence of carryover effects across blocks, participants also engaged in a counting task at the conclusion of each block. We conducted ROI analyses of bilateral amygdalae to compare activation patterns during relevant trials of the Social Evaluation Task (negative immerse > neutral immerse) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | 0.04 (0.23) | -0.01 (0.31)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. An ROI mask was generated from left and right amygdala of the AAL1.V4 atlas. First-level contrast estimates (negative immerse > neutral immerse) for each voxel within the ROI were averaged with MarsBaR to produce a single value for each person. A two-sample t-test was conducted in R to test for differences across intervention groups (mindset vs control); p = 0.265, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(146) = -1.12

8. Primary Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Amygdala Activation- Go/No-go Task
Description: The Socioemotional Go/No-go Task examines inhibitory control in the presence of socioemotional distractors. Participants were presented with a socially aversive image, or neutral image for 300ms. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond quickly to every letter except an infrequent nontarget letter. We conducted ROI analyses of bilateral amygdalae to compare activation patterns of emotion reactivity during relevant trials of the Socioemotional Go/No-go Task (negative > neutral) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 75
BOLD signal change | 0.49 (0.45) | 0.49 (0.54)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. An ROI mask was generated from left and right amygdala of the AAL1.V4 atlas. First-level contrast estimates (negative > neutral) for each voxel within the ROI were averaged with MarsBaR to produce a single value for each person. A two-sample t-test was conducted in R to test for differences across intervention groups (mindset vs control); p = 0.96, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(145) = -0.53

9. Primary Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Frontal Parietal Network-Amygdala Connectivity- Social Evaluation Task
Description: The Social Evaluation Task (SET) examines emotion reactivity and regulation with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative condition), praise (positive condition) or neutral statements (neutral condition). Participants were asked to imagine the person was either an actor practicing lines (reframe condition), or a close friend (immerse condition). Participants were subsequently asked to rate how they felt on a 5 item Likert scale from "Very Good" to "Very Bad". To reduce the influence of carryover effects across blocks, participants also engaged in a counting task at the conclusion of each block. Psychophysiological interaction (PPI) analysis was conducted in SPM12 to examine task-dependent changes in connectivity between amygdalae and frontoparietal network (FPN) during relevant trials (negative reframe > negative immerse) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | 0.01 (0.41) | -0.01 (0.33)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were preprocessed in fMRIprep. Separate right/left amygdala seeds were defined with the AAL1 atlas. Interaction regressors were created between seeds and task conditions. Average contrast estimates for interaction terms of relevant trials (negative reframe > negative immerse) were extracted with MarsBaR from 15 ROIs in the FPN of a modified Schaefer atlas and the 30 values averaged. A two-sample t-test was conducted in R to compare average connectivity between groups (mindset vs control); p = 0.76, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(146) = -.3047

10. Primary Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Frontal Parietal Network-Amygdala Connectivity- Go/No-go Task
Description: The Socioemotional Go/No-go Task examines inhibitory control in the presence of socioemotional distractors. Participants were presented with a socially aversive image, or neutral image for 300ms. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond quickly to every letter except an infrequent nontarget letter. Psychophysiological interaction (PPI) analysis was conducted in SPM12 to examine task-dependent changes in connectivity between amygdalae and frontoparietal network (FPN) during relevant trials of the Socioemotional Go/No-go Task (negative > neutral) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | -0.17 (0.61) | 0.01 (0.48)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were preprocessed in fMRIprep. Separate right/left amygdala seeds were defined with the AAL1 atlas. Interaction regressors were created between seeds and task conditions. Average contrast estimates for interaction terms of relevant trials (negative > neutral) were extracted with MarsBaR from 15 ROIs in the FPN of a modified Schaefer atlas and the 30 values averaged. A two-sample t-test was conducted in R to compare average connectivity between groups (mindset vs control); p = .048, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(145) = 1.998, p = .048

11. Primary Outcome: Mean Change on Self-Reported State Negative Affect
Description: Before (Pre-trier negative affect) and after (Post-trier negative affect) completing the Trier Social Stress Test (TSST) at baseline, participants completed ratings of negative emotions (10 items), modified from another affect measure (Owens et al., 2019), to test the efficacy of the TSST. Participants rated their emotions on a 100-point scale (0 = Not at All to 100 = Extremely) to indicate the extent they were feeling a negative emotion at that particular moment. Scores were computed as the mean of the items, with higher scores reflecting higher levels of negative emotions. In this analysis, we compared mean change scores across the two conditions (mindset and control).
Time Frame: Pre-Trier vs. Post-Trier: baseline
Population: Six participants declined participation on this task.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 77 | 80
score on a scale
  Pre-trier negative affect | 6.93 (9.66) | 8.00 (8.63)
  Post-trier negative affect | 15.05 (14.83) | 16.51 (14.35)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.833, ANOVA; degrees of freedom =1

12. Primary Outcome: Mean Difference on Self-Reported Affect on Social Evaluation Task
Description: The Social Evaluation Task examines emotion reactivity and regulation in the context of social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative immerse or reframe), praise (positive immerse or reframe), or neutral statements (neutral immerse). In immerse trials, participants imagined that the person was a close friend. During the reframe trials, participants imagined that the person was an actor. After each trial, participants rated how they felt from 1 (Very Good) to 5 (Very Bad). Means of each condition were computed with higher scores indicating more negative emotions. In this analysis, we compared mean difference between criticism and praise vs. neutral trials across the two conditions (mindset and control) for the Social Evaluation Task
Time Frame: Post Mindset Manipulation: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 74 | 76
units on a scale
  negative immerse | 4.34 (0.51) | 4.28 (0.63)
  positive immerse | 1.61 (0.60) | 1.61 (0.58)
  negative reframe | 3.49 (0.51) | 3.45 (0.67)
  positive reframe | 2.39 (0.64) | 2.32 (0.60)
  neutral immerse | 2.90 (0.33) | 2.87 (0.43)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group effect (Growth Mindset vs. Brain Education) across self-reported affect on the SET task. This is a test of between-subjects effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.321, ANOVA; degrees of freedom = 1

13. Secondary Outcome: Mean Change From Baseline to 2 Months in Emotion Mindset Scale Scores
Description: Participants completed a six-item fixed emotion mindset measure (EMS-fixed) measure, prior to (pre-induction EMS) the induction lessons and again at at 2-month follow-up. Items were drawn from the Implicit Theories of Emotion Scale (Tamir et al., 2007) and the Emotion Mindset Scale (EMS; Livingstone, 2013). Participants rated each item on a 6-point scale (1 = Strongly Disagree to 6 =Strongly Agree). Means were computed for these items, with higher scores representing a higher fixed emotion mindset mindset. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=6 High=better outcome
Time Frame: At baseline and in approximately 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 81 | 82
score on a scale
  pre-induction child fixed emotion mindset | 3.03 (0.96) | 3.03 (0.92)
  post-induction child fixed emotion mindset (2months) | 2.74 (1.00) | 3.17 (1.01)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) for fixed emotion mindset scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.002, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on fixed emotion mindset scores from time 1 to time 2. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.005, ANCOVA; degrees of freedom = 1

14. Secondary Outcome: Mean Change From Baseline to 4 Months in Emotion Mindset Scores
Description: Participants completed a six-item fixed emotion mindset measure (EMS-fixed) measure, prior to (pre-induction EMS) the induction lessons and again at at 4-month follow-up. Items were drawn from the Implicit Theories of Emotion Scale (Tamir et al., 2007) and the Emotion Mindset Scale (EMS; Livingstone, 2013). Participants rated each item on a 6-point scale (1 = Strongly Disagree to 6 =Strongly Agree). Means were computed for these items, with higher scores representing a higher fixed emotion mindset mindset. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=6 High=better outcome
Time Frame: At baseline and in approximately 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 81 | 82
score on a scale
  pre-induction child fixed emotion mindset | 3.03 (0.96) | 3.03 (0.92)
  post-induction child fixed emotion mindset (4months) | 2.80 (0.98) | 3.11 (0.92)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on fixed emotion mindset scores from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = .033, ANOVA; degrees of freedom = 1

15. Secondary Outcome: Mean Change From Baseline to 2 Months in Emotional Self-efficacy Scale Scores (Measure Beliefs About Ability to Control Emotions)
Description: Participants completed a measure assessing their perceived ability to manage emotions prior to the induction and again at a 2-month follow-up. Items were derived from the using and managing your own emotions subscale of the Youth-Emotional Self-efficacy Scale (5 items; Qualter et al., 2015). Participants rated the items on a 5-point Likert scale (1 = Disagree Strongly to 5 = Agree Strongly). Scores were computed as the mean of the items, with higher scores indicating greater emotion regulation self-efficacy. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome.
Time Frame: At baseline and in approximately 2 months
Population: Because only 69 participants in the growth mindset condition and 66 participants in the brain education completed the follow-up at 2-months, these analyses included only the same 69 and 66 participants who also completed the measure at baseline. Thus, the sample at baseline for pre-induction emotional self-efficacy is smaller in these analyses and the mean is different for baseline than it was initially at baseline because it includes a smaller portion of the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 69 | 66
score on a scale
  pre-induction emotional self-efficacy | 3.64 (0.68) | 3.38 (0.93)
  post-induction emotional self-efficacy (2months) | 3.55 (0.76) | 3.40 (0.93)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — Threshold for statistical significance was p = 0.05; p = 0.403, ANOVA; degrees of freedom =1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy scores from time 1 to time 2. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.190, ANCOVA; degrees of freedom = 1

16. Secondary Outcome: Mean Change From Baseline to 4 Months in Emotional Self-efficacy Scale Scores (Measure Beliefs About Ability to Control Emotions)
Description: Participants completed a measure assessing their perceived ability to manage emotions prior to the induction and again at a 4-month follow-up. Items were derived from the using and managing your own emotions subscale of the Youth-Emotional Self-efficacy Scale (5 items; Qualter et al., 2015). Participants rated the items on a 5-point Likert scale (1 = Disagree Strongly to 5 = Agree Strongly). Scores were computed as the mean of the items, with higher scores indicating greater emotion regulation self-efficacy. Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome.
Time Frame: At baseline and in approximately 4 months
Population: Because only 70 participants in the growth mindset condition and 70 participants in the brain education completed the follow-up at 4-months, the number analyzed includes only the same 70 and 70 participants who also completed the measure at baseline. Thus, the sample at baseline for pre-induction emotional self-efficacy is smaller in these analyses and the mean is different for baseline than it was initially at baseline because it includes a smaller portion of the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 70 | 70
score on a scale
  pre-induction emotional self-efficacy | 3.64 (0.67) | 3.37 (0.91)
  post-induction emotional self-efficacy (4months) | 3.63 (0.69) | 3.39 (0.94)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy scores from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.784, ANOVA — degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy scores from time 1 to time 3. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.586, ANCOVA; degrees of freedom =1

17. Secondary Outcome: Mean Change From Baseline to 2 Months in Emotional Self-efficacy Vignettes Scores
Description: To assess emotion regulation self-efficacy participants completed a self-efficacy measure adapted from Tamir and colleagues (2007). Prior to the induction and again. at a 2-month follow-up, participants were asked to rate 12 emotion-eliciting events drawn from daily life. Three scenarios were adapted from the Tamir self-efficacy measure (Tamir et al. 2007. Participants rated how confident they were in their ability to control their emotions in each scenario on a 5-point scale (1 = Not at All to 5 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting greater self-efficacy.Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome
Time Frame: At baseline and in approximately 2 months
Population: Because only 69 participants in the growth mindset condition and 66 participants in the brain education completed the follow-up at 2-months, the number analyzed includes only the same 69 and 66 participants who also completed the measure at baseline. Thus, the sample at baseline for pre-induction emotional self-efficacy vignettes is smaller in these analyses and the mean is different for baseline than it was initially at baseline because it includes a smaller portion of the sample.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 69 | 66
units on a scale
  pre-induction emotional self-efficacy vignette score | 2.95 (0.61) | 2.70 (0.65)
  post-induction emotional self-efficacy vignette score (2months) | 2.93 (0.69) | 2.69 (0.66)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy vignette scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.916, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy vignette scores from time 1 to time 2. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.343, ANCOVA; degrees of freedom =1

18. Secondary Outcome: Mean Change From Baseline to 4 Months in Emotional Self-efficacy Vignettes Scores
Description: To assess emotion regulation self-efficacy participants completed a self-efficacy measure adapted from Tamir and colleagues (2007). Prior to the induction and again at a 4-month follow-up, participants were asked to rate 12 emotion-eliciting events drawn from daily life. Three scenarios were adapted from the Tamir self-efficacy measure (Tamir et al. 2007. Participants rated how confident they were in their ability to control their emotions in each scenario on a 5-point scale (1 = Not at All to 5 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting greater self-efficacy.Will compare mean change scores across the two conditions (mindset and control) Minimum=1 Maximum=5 High=better outcome
Time Frame: At baseline and in approximately 4 months
Population: Because only 69 participants in the growth mindset condition and 69 participants in the brain education completed the follow-up at 4-months, the number analyzed includes only the same 70 and 70 participants who also completed the measure at baseline. Thus, the sample at baseline for pre-induction emotional self-efficacy vignettes is smaller in these analyses and the mean is different for baseline than it was initially at baseline because it includes a smaller portion of the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 69 | 70
score on a scale
  pre-induction emotional self-efficacy vignettes score | 2.95 (0.59) | 2.71 (0.62)
  post-induction emotional self-efficacy vignettes score (4months) | 3.19 (0.68) | 2.74 (0.60)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy vignette scores from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.048, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on emotional self-efficacy vignette scores from time 1 to time 3. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lesson was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.153, ANCOVA; degrees of freedom = 1

19. Secondary Outcome: Mean Change From Baseline to 2 Months in Self-Reported Emotion Regulation Strategies Scores
Description: To assess emotion (dys)regulation, participants completed a novel 44-item emotion regulation measure at baseline and again at a 2-month follow-up. Items were rated on a 5-point scale (1 = Not at All to 5 = Very Much). Factor analyses yielded three emotion regulation strategies factors- proactive engagement, involuntary dysregulation, and disengagement. Scores were computed as the mean of the items on each factor (1 = Not at All to 5 = Very Much), with higher scores reflecting higher levels of type of response. Higher scores on proactive engagement are considered adaptive and higher scores on involuntary dysregulation are maladaptive.
  Will compare mean change scores across the two conditions (mindset and control)
Time Frame: At baseline and in approximately 2 months
Population: Some participants did not complete all of the items and thus their emotion regulation strategies factors could not be calculated. Because only 72-73 participants in the growth mindset condition and 70-71 participants in the brain education completed the follow-up at 2-months (some participants filled out half the measure), the number analyzed includes only the same 72-73 and 70-71 participants who also completed the measure at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 73 | 71
score on a scale
  Pre-induction ERD proactive engagement: number analyzed (Participants) | 73 | 70
  Pre-induction ERD proactive engagement | 2.97 (0.80) | 2.69 (0.78)
  Post-induction ERD proactive engagement (2Months): number analyzed (Participants) | 73 | 70
  Post-induction ERD proactive engagement (2Months) | 3.07 (0.74) | 2.85 (0.75)
  Pre-induction ERD involuntary dysregulation: number analyzed (Participants) | 72 | 71
  Pre-induction ERD involuntary dysregulation | 2.40 (0.63) | 2.45 (0.77)
  Post-induction ERD involuntary dysregulation (2months): number analyzed (Participants) | 72 | 71
  Post-induction ERD involuntary dysregulation (2months) | 2.44 (0.68) | 2.68 (0.79)
  Pre-induction ERD disengagement | 3.28 (0.62) | 3.05 (0.73)
  Post-induction ERD disengagement (2months) | 3.30 (0.66) | 3.17 (0.68)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD proactive engagement scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.566, ANOVA; degrees of freedom =1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD involuntary dysregulation scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.048, ANOVA; degrees of freedom = 1
Statistical Analysis 3: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD involuntary dysregulation scores from time 1 to time 2. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.266, ANCOVA; degrees of freedom =1
Statistical Analysis 4: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD disengagement scores from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.402, ANOVA; degrees of freedom =1

20. Secondary Outcome: Mean Change From Baseline to 4 Months in Self-Reported Emotion Regulation Strategies Scores
Description: To assess emotion (dys)regulation, participants completed a novel 44-item emotion regulation measure at baseline and again at a 4-month follow-up. Items were rated on a 5-point scale (1 = Not at All to 5 = Very Much). Factor analyses yielded three emotion regulation strategies factors- proactive engagement, involuntary dysregulation, and disengagement. Scores were computed as the mean of the items on each factor (1 = Not at All to 5 = Very Much), with higher scores reflecting higher levels of type of response. Higher scores on proactive engagement are considered adaptive and higher scores on involuntary dysregulation are maladaptive.
  Will compare mean change scores across the two conditions (mindset and control) Will compare mean change scores across the two conditions (mindset and control)
Time Frame: At baseline and in approximately 4 months
Population: Some participants did not complete all of the items and thus their emotion regulation strategies factors could not be calculated. Because only 71-72 participants in the growth mindset condition (some participants filled out half the measure) and 74 participants in the brain education completed the follow-up at 4-months, the number analyzed includes only the same 71-72 and 74 participants who also completed the measure at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 74
score on a scale
  Pre-induction ERD proactive engagement | 2.96 (0.79) | 2.73 (0.78)
  Post-induction ERD proactive engagement (4months) | 3.12 (0.72) | 2.78 (0.74)
  Pre-induction ERD involuntary dysregulation | 2.42 (0.64) | 2.49 (0.78)
  Post-induction ERD involuntary dysregulation (4months) | 2.47 (0.79) | 2.64 (0.83)
  Pre-induction ERD disengagement: number analyzed (Participants) | 71 | 74
  Pre-induction ERD disengagement | 3.23 (0.68) | 2.99 (0.71)
  Post-induction ERD disengagement (4months): number analyzed (Participants) | 71 | 74
  Post-induction ERD disengagement (4months) | 3.28 (0.66) | 3.15 (0.75)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD proactive engagement from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.363, ANOVA; degrees of freedom =1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD involuntary dysregulation scores from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.363, ANOVA; degrees of freedom = 1
Statistical Analysis 3: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD involuntary dysregulation scores from time 1 to time 3. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.583, ANCOVA; degrees of freedom = 1
Statistical Analysis 4: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD disengagement scores from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.379, ANOVA; degrees of freedom = 1
Statistical Analysis 5: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (pre-manipulation and post-manipulation) on ERD disengagement scores from time 1 to time 3. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.246, ANCOVA; degrees of freedom = 1

21. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Cingulo-Opercular Network Activation- Social Evaluation Task
Description: The Social Evaluation Task (SET) examines emotion reactivity and regulation with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative condition), praise (positive condition) or neutral statements (neutral condition). Participants were asked to imagine the person was either an actor practicing lines (reframe condition), or a close friend (immerse condition). Participants were subsequently asked to rate how they felt on a 5 item Likert scale from "Very Good" to "Very Bad". To reduce the influence of carryover effects across blocks, participants also engaged in a counting task at the conclusion of each block. We conducted ROI analyses of the cingulo-opercular network (CON) to compare activation patterns of emotion reactivity during relevant trials (negative reframe > negative immerse) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | -0.07 (0.41) | -0.02 (0.37)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. 12 ROI masks were generated from the CON network of a modified Schaefer atlas. First-level contrast estimates (negative reframe > negative immerse) for each voxel within each ROI were averaged with MarsBaR to produce 12 values for each person. These were then averaged to produce a single value each.A two-sample t-test was conducted in R to test for differences across intervention groups (mindset vs control); p = 0.455, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(146) = .75

22. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Cingulo-Opercular Network Activation- Go/No go Task
Description: The Socioemotional Go/No-go Task examines inhibitory control in the presence of socioemotional distractors. Participants were presented with a socially aversive image, or neutral image for 300ms. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond quickly to every letter except an infrequent nontarget letter. We conducted ROI analyses of the cingulo-opercular network (CON) to compare activation patterns during relevant trials of the Socioemotional Go/No-go Task (negative > neutral) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 75
BOLD signal change | -0.11 (0.62) | -0.02 (0.68)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. 12 ROI masks were generated from the CON network of a modified Schaefer atlas. First-level contrast estimates (negative > neutral) for each voxel within each ROI were averaged with MarsBaR to produce 12 values for each person. These were subsequently averaged to produce a single value per person. A two-sample t-test was conducted in R to test for differences across intervention groups (mindset vs control); p = 0.43, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(145) = 0.80

23. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Cingulo-Opercular Network Activation- Resting State
Description: We conducted ROI analyses of the cingulo-opercular network (CON) to explore difference in mean intrinsic neural activity across experimental conditions (mindset vs control). Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. 12 ROI masks were generated from the CON network of a modified Schaefer atlas.
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Error); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 70 | 74
BOLD signal change | -0.0000003502 (0.00002200) | 0.000003274 (0.00001911)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — BOLD signals were spatially averaged within ROIs to produce a single time series for each ROI. Timeseries were averaged to produce a single value representing each ROI's mean activity. Values for each ROI were then averaged to produce a single value per person representing mean network activity. These values were then submitted to a two-sample t-test to test for differences across intervention groups (mindset vs control); p = 0.29, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(142) = -1.057

24. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal Cingulo-Opercular Network-Amygdala Connectivity- Social Evaluation Task
Description: The Social Evaluation Task (SET) examines emotion reactivity and regulation with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative condition), praise (positive condition) or neutral statements (neutral condition). Participants were asked to imagine the person was either an actor practicing lines (reframe condition), or a close friend (immerse condition). Participants were subsequently asked to rate how they felt on a 5 item Likert scale from "Very Good" to "Very Bad". To reduce the influence of carryover effects across blocks, participants also engaged in a counting task at the conclusion of each block. Psychophysiological interaction (PPI) analysis was conducted in SPM12 to examine task-dependent changes in connectivity between amygdalae and cingulo-opercular network (CON) during relevant trials (negative reframe > negative immerse) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | -0.005 (0.40) | 0.004 (0.34)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were preprocessed in fMRIprep. Separate right/left amygdala seeds were defined with the AAL1 atlas. Interaction regressors were created between seeds and task conditions. Average contrast estimates for interaction terms of relevant trials (negative reframe > negative immerse) were extracted with MarsBaR from 12 ROIs in the CON of a modified Schaefer atlas and the 24 values averaged. A two-sample t-test was conducted in R to compare average connectivity between groups (mindset vs control); p = 0.88, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(146) = 0.148

25. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal for Cingulo-Opercular Network-Amygdala Connectivity- Go/no go Task
Description: The Socioemotional Go/No-go Task examines inhibitory control in the presence of socioemotional distractors. Participants were presented with a socially aversive image, or neutral image for 300ms. After the image, a white box with a black letter was superimposed on the image for 500 ms. Participants were instructed to respond quickly to every letter except an infrequent nontarget letter. Psychophysiological interaction (PPI) analysis was conducted in SPM12 to examine task-dependent changes in connectivity between amygdalae and cingulo-opercular network (CON) during relevant trials (negative > neutral) across experimental conditions (mindset vs control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change | -0.12 (0.60) | 0.03 (0.49)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — Data were preprocessed in fMRIprep. Separate right/left amygdala seeds were defined with the AAL1 atlas. Interaction regressors were created between seeds and task conditions. Average contrast estimates for interaction terms of relevant trials (negative > neutral) were extracted with MarsBaR from 12 ROIs in the CON of a modified Schaefer atlas and the 24 values averaged. A two-sample t-test was conducted in R to compare average connectivity between groups (mindset vs control); p = .11, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(145) = 1.631

26. Other Pre Specified Outcome: Mean Difference in Parameter Estimates of BOLD Signal Cingulo-Opercular Network-Amygdala Connectivity- Resting State
Description: Data were collected using a Siemens Prisma MRI 3T scanner and preprocessed with fMRIprep. We conducted connectivity analysis between the cingulo-opercular network (CON) and bilateral amygdala to explore difference in mean intrinsic CON-amygdala neural connectivity across experimental conditions (mindset vs control). 12 ROI masks were generated from the CON network of a modified Schaefer atlas. Separate right/left amygdala seeds were defined with the AAL1 atlas.
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 70 | 74
BOLD signal change | 0.20 (0.12) | 0.20 (0.10)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; A two-sample t-test was conducted to compare average connectivity (between the amygdala and the CON network) during resting state between the mindset and control groups; Test type: Superiority — BOLD signals were spatially averaged within ROIs to produce a single time series for each ROI. Pearson correlations were calculated between each mean BOLD signal in the CON and each amygdala ROI to produce 24 connectivity values. These were averaged to produce a single value representing the strength of coupling of the CON network to the amygdala for each participant. These values were then submitted to a two-sample t-test to test for differences across intervention groups (mindset vs control); p = 0.92, t-test, 2 sided — The threshold for statistical significance was p < 0.05; t(142) = 0.101

27. Other Pre Specified Outcome: Group Differences in Parameter Estimates of BOLD Signal for Whole-Brain Analyses- Social Evaluation Task
Description: The Social Evaluation Task (SET) examines emotion reactivity and regulation with social stimuli. Stimuli consisted of video clips with actors expressing criticism (negative condition), praise (positive condition) or neutral statements (neutral condition). Participants were asked to imagine the person was either an actor practicing lines (reframe condition), or a close friend (immerse condition). Participants were subsequently asked to rate how they felt on a 5 item Likert scale from "Very Good" to "Very Bad". To reduce the influence of carryover effects across blocks, participants also engaged in a counting task at the conclusion of each block. We conducted exploratory whole-brain voxelwise analyses in SPM12 to compare activation patterns during relevant trials of the Social Evaluation Task (negative immerse > neutral immerse and negative reframe > negative immerse) across experimental conditions (mindset > control).
Time Frame: Post Mindset Manipulation: baseline
Population: Some participants declined participation in these tasks and other data was lost due to technological error.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 76
BOLD signal change
  Anterior Cingulate/Medial Frontal Gyrus | 0.37167 (0.49233) | 0.01202 (0.51865)
  Middle Frontal Gyrus (Left) | 0.17254 (0.30488) | -0.07882 (0.33388)
  Posterior Cingulate/Cingulate | 0.16448 (0.37390) | -0.09570 (0.45070)
  Middle Temporal Gyrus (Left) | 0.08163 (0.54079) | -0.33910 (0.60712)
  Middle Frontal Gyrus (Right) | 0.13315 (0.35573) | -0.13705 (0.39000)
  Superior/Middle Temporal Gyrus (Right) | 0.29583 (0.49264) | -0.06817 (0.56753)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; Test type: Other — Data were preprocessed in fMRIprep. A first-level contrast estimate of interest (negative immerse > neutral immerse) was submitted to a second-level t-test for group-level differences across experimental conditions (mindset > control). Monte Carlo simulations using 3dClustSim in AFNI controlled cluster-level family-wise error rate at p < 0.001 with a cluster-defining threshold of p < 0.005. The WFU PickAtlas via xjview was used to determine anatomical localization for surviving clusters; p = .0000222, t-test, 2 sided — Reported result for cluster localized in the Superior/Middle Temporal Gyrus (Right). FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — [test comment as in outcome 27, analysis 1]; p = .0000117, t-test, 2 sided — Reported result for cluster localized in the Middle Temporal Gyrus (Left). FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 3: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — [test comment as in outcome 27, analysis 1]; p = .000000000, t-test, 2 sided — Reported result for cluster localized in the Anterior Cingulate/Medial Frontal Gyrus. FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 4: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — [test comment as in outcome 27, analysis 1]; p = .0000186, t-test, 2 sided — Reported result for cluster localized in the Middle Frontal Gyrus (Right). FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 5: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — [test comment as in outcome 27, analysis 1]; p = .000000000, t-test, 2 sided — Reported result for cluster localized in the Middle Frontal Gyrus (Left). FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 6: Comparison: Growth Mindset vs Brain Education; Test type: Superiority — [test comment as in outcome 27, analysis 1]; p = .0000161, t-test, 2 sided — Reported result for cluster localized in the Posterior Cingulate/Cingulate. FWE-corrected p-value is reported. pvoxel-level < .005, pcluster-level < .001. Cluster extent = 278 voxels
Statistical Analysis 7: Comparison: Growth Mindset vs Brain Education; Test type: Other — Data were preprocessed in fMRIprep. A first-level contrast estimate of interest (negative reframe > negative immerse) was submitted to a second-level t-test for group-level differences across experimental conditions (mindset > control). Monte Carlo simulations using 3dClustSim in AFNI controlled cluster-level family-wise error rate at p < 0.001 with a cluster-defining threshold of p < 0.005; p > .001, t-test, 2 sided — pvoxel-level < .005, pcluster-level < .001. Cluster extent = 298 voxels

28. Other Pre Specified Outcome: Mean Change From Baseline to 2 Months in Depressive Symptoms Scores
Description: Participants completed the short form of the Mood and Feelings Questionnaire (SMFQ; Angold et al., 1995) to assess depressive symptoms (13 items) at baseline and again at a 2-month follow-up. The original version was modified (Liang & Eley, 2005) to provide a 4-point response format (1 = Not at All, 2 = A Little Bit, 3 = Pretty Much, 4 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting higher levels of depressive symptoms.
  Will compare mean change scores across the two conditions (mindset and control) at baseline and the two month follow-up.
Time Frame: At baseline and in approximately 2 months
Population: Because only 71 participants in the growth mindset condition and 70 participants in the brain education completed the follow-up at 2-months, the number analyzed includes only the same 71 and 70 participants who completed the measure at baseline and follow-up. The number of participants and means are different at baseline because these include a smaller set of the sample than initially at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 71 | 70
score on a scale
  Baseline depression (SMFQ) | 1.81 (0.69) | 1.84 (0.67)
  Follow-up depression (SMFQ; 2months) | 1.91 (0.74) | 2.00 (0.74)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (baseline and follow-up) on depression levels from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.560, ANOVA; degrees of freedom = 1

29. Other Pre Specified Outcome: Mean Change From Baseline to 4 Months in Depressive Symptoms Scores
Description: Participants completed the short form of the Mood and Feelings Questionnaire (SMFQ; Angold et al., 1995) to assess depressive symptoms (13 items) at baseline and again at a 4-month follow-up. The original version was modified (Liang & Eley, 2005) to provide a 4-point response format (1 = Not at All, 2 = A Little Bit, 3 = Pretty Much, 4 = Very Much). Scores were computed as the mean of the items, with higher scores reflecting higher levels of depressive symptoms.
  Will compare mean change scores across the two conditions (mindset and control) at baseline and the four-month follow-up.
Time Frame: At baseline and in approximately 4 months
Population: Because only 71 participants in the growth mindset condition and 72 participants in the brain education completed the follow-up at 4-months, the number analyzed includes only the same 71 and 72 participants who completed the measure at baseline and follow-up. The number of participants and means are different at baseline because these include a smaller set of the sample than initially at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 71 | 72
score on a scale
  Baseline depression (SMFQ) | 1.81 (0.68) | 1.82 (0.67)
  Follow-up depression (SMFQ; 4months) | 1.94 (0.72) | 2.05 (0.82)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (baseline and follow-up) on depression levels from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.327, ANOVA; degrees of freedom = 1

30. Other Pre Specified Outcome: Mean Change From Baseline to 2 Months in Anxiety Symptoms Scores
Description: Participants completed the Revised Child Manifest Anxiety Scale (RCMAS; Reynolds & Richmond, 1985) at baseline and again at a 2-month follow-up. The RCMAS includes 28 items assessing anxiety symptoms (e.g., "I often worry about something bad happening to me.") rated on a dichotomous scale (0 = No, 1 = Yes). Total anxiety scores were created by taking the sum of the items, with higher scores reflecting higher levels of anxiety. The RCMAS shows strong internal consistency (Reynolds & Richmond, 1978) and test-retest reliability (Wisniewski et al., 1987). Will compare mean change scores across the two conditions (mindset and control)
Time Frame: At baseline and in approximately 2 months
Population: Because only 72 participants in the growth mindset condition and 69 participants in the brain education completed the follow-up at 2-months, the number analyzed includes only the same 72 and 69 participants who completed the measure at baseline and follow-up. The number of participants and means are different at baseline because these include a smaller set of the sample than initially at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 72 | 69
score on a scale
  Baseline anxiety (RCMAS) | 13.04 (5.98) | 13.98 (6.37)
  Follow-up anxiety (RCMAS; 2months) | 13.60 (7.17) | 15.21 (7.55)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (baseline and follow-up) on anxiety levels from time 1 to time 2. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.439, ANOVA; degrees of freedom = 1
Statistical Analysis 2: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (baseline and follow-up) on anxiety levels from time 1 to time 2. This is a test of between by within-subjects interaction effect. Clarity of the psycho-educational lessons was included as a covariate; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.545, ANCOVA; degrees of freedom = 1

31. Other Pre Specified Outcome: Mean Change From Baseline to 4 Months in Anxiety Symptoms Scores
Description: Participants completed the Revised Child Manifest Anxiety Scale (RCMAS; Reynolds & Richmond, 1985) at baseline and again at a 4-month follow-up. The RCMAS includes 28 items assessing anxiety symptoms (e.g., "I often worry about something bad happening to me.") rated on a dichotomous scale (0 = No, 1 = Yes). Total anxiety scores were created by taking the sum of the items, with higher scores reflecting higher levels of anxiety. The RCMAS shows strong internal consistency (Reynolds & Richmond, 1978) and test-retest reliability (Wisniewski et al., 1987). Will compare mean change scores across the two conditions (mindset and control). Will compare mean change scores across the two conditions (mindset and control)
Time Frame: At baseline and in approximately 4 months
Population: Because only 70 participants in the growth mindset condition and 73 participants in the brain education completed the follow-up at 4-months, the number analyzed includes only the same 70 and 73 participants who completed the measure at baseline and follow-up. The number of participants and means are different at baseline because these include a smaller set of the sample than initially at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Growth Mindset | Brain Education
Number analyzed (Participants) | 70 | 73
score on a scale
  Baseline anxiety (RCMAS) | 13.50 (6.09) | 13.60 (6.30)
  Follow-up anxiety (RCMAS; 4months) | 13.53 (7.36) | 13.92 (7.03)
Statistical Analysis 1: Comparison: Growth Mindset vs Brain Education; We are reporting the p-value for the group (Growth Mindset vs. Brain Education) by time effect (baseline and follow-up) on anxiety levels from time 1 to time 3. This is a test of between by within-subjects interaction effect; Test type: Superiority — The threshold for statistical significance was p = 0.05; p = 0.740, ANOVA; degrees of freedom = 1

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Arm/Group | Growth Mindset | Brain Education
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03978871/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03978871/SAP_001.pdf
  • Informed Consent Form: Parent Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03978871/ICF_002.pdf
  • Informed Consent Form: Child Assent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03978871/ICF_003.pdf